CLINICAL TRIAL: NCT02087566
Title: Single-Dose Linezolid Pharmacokinetics In Critically Ill Patients With Impaired Renal Function Especially Chronic Haemodialysis Patients
Brief Title: Linezolid Pharmacokinetics In Patients With Impaired Renal Function (PPT6)
Acronym: LZDPPT6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sally Helmy, PhD, CPHQ, Faculty of Pharmacy-Damanhour University, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: LZDPPT6
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Renal Failure; Impaired Renal Function
Keywords: Linezolid; Pharmacokinetics; Haemodialysis; Dosing adjustment; Eligible subjects were classified into three groups depending on their 24-h urinary creatinine clearance (CLcr) values or HD status.; Group 1, included 6 healthy subjects with normal renal function (CLcr ˃80 ml/min);; Group 2, included 6 patients with acute renal failure (RF) (30˂CLcr˂80 ml/mine);; Group 3, included 6 patients on long term haemodialysis (minimum period of dialysis was 40 month while maximum period were 130 month)
MeSH Terms: conditions — Renal Insufficiency | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Administration of linezolid to 6 healthy volunteers (Other): Administration of linezolid to 6 healthy volunteers {six healthy subjects with normal renal function (CLcr ˃80 ml/min)}
  Interventions: Drug: 600 mg linezolid
- Administration of linezolid to 6 acute renal failure patients (Other): Administration of linezolid to 6 acute renal failure patients {(six patients with acute renal failure (RF) (30˂CLcr˂80 ml/mine)}
  Interventions: Drug: 600 mg linezolid
- Administration of linezolid to 6 ESRD patients (Other): Administration of linezolid to 6 end-stage renal disease (ESRD) patients during an intra-dialytic period (on-dialysis): 6 patients on long term HD (minimum period of dialysis was 40 month while maximum period were 130 month) with an ideal body weight of >60 kg (calculated as {height (cm) -100}×0.9) and a body mass index between 20 and 26 kg/m2 (calculated as {weight (kg)/height (m2)}).
  Interventions: Drug: 600 mg linezolid

INTERVENTIONS:
Drug: 600 mg linezolid

SUMMARY:
Renal failure patients were treated with linezolid (LZD) for proven or suspected infections by multiresistant Gram-positive cocci. The aim of this study is to determine if dose adjustment of LZD is needed as a function of renal impairment or not, especially that a significant component of LZD is eliminated unchanged in urine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with normal renal function (CLcr ˃80 ml/min);
* Patients with acute renal failure (RF) (30˂CLcr˂80 ml/mine)
* Patients on long term HD with an ideal body weight of >60 kg and a body mass index between 20 and 26 kg/m2
* Passed all the screening parameters
* Free of any drug exposure known to interfere with the pharmacokinetics or assay of linezolid for at least 10 days prior to the study
* Able to communicate effectively with study personnel, be literate, and able to give consent.

Exclusion Criteria:

Had a history of clinically significant organ dysfunction other than renal disease or those diseases associated with renal disease (as in case of acute RF or ESRD patients) Had physical examination or laboratory test results outside the inclusion such as; sitting systolic BP (SBP) of >140 or <100 mmHg, diastolic BP (DBP) > 90 or <60mm Hg (as in case of healthy volunteers and acute RF patients), or a pulse rate of > 95 or < 50 beats/min at screening; history of orthostatic hypotension; history of serious intolerance, allergy or sensitivity to linezolid ; history of blood dyscrasias; history of alcohol, smoking, or drug abuse; donation of blood during the 8 weeks prior to the study or plans to donate blood during or within 8 weeks of completing the study; unable to tolerate vein puncture and multiple blood samplings; any surgical/medical condition that might alter the absorption, distribution, metabolism, excretion of linezolid ; or can't follow instructions, according to the investigator's opinion.

-

Ages: 22 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Tolerability | Participants will be followed for the duration of study, an expected average of 6 weeks.
  Tolerability was assessed based on changes in vital signs (temperature, blood pressure, pulse, and heart rate), measured before dosing in each period and approximately every 4 hours thereafter, and laboratory tests (hematology, biochemistry, liver function, and urinalysis), and performed at baseline and at the end of the study. In addition, a physician questioned volunteers about any adverse events occurring during the study, addressed them as necessary, and recorded them on the appropriate form. This physician was not blinded to treatment, but had no involvement in the study.